CLINICAL TRIAL: NCT03193619
Title: A Prospective, Multi-Center, Single-Arm, Real-World Study Assessing the Clinical Use of the Bard® UltraScore™ Focused Force PTA Balloon
Brief Title: Real World Registry Assessing the Clinical Use of the Bard UltraScore Forced Focus PTA Balloon
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: BPV-16-001
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases; Arterial Occlusive Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- PTA-UltraScore Focused Force PTA balloon: Treatment with the UltraScore Focused Force PTA balloon will be per the investigational site's standard of care and adhering to the IFU.
  Interventions: Device: PTA (UltraScore Focused Force PTA Balloon)

INTERVENTIONS:
Device: PTA (UltraScore Focused Force PTA Balloon) — Percutaneous Transluminal Angioplasty (PTA) will involve the insertion of a catheter into one of the femoral arteries. Once the catheter is in place, a tiny balloon on the end of the catheter will be inflated to press against the narrowing (or blockage) in the artery to try to open the blockage, and allow more blood to flow through the artery. The balloon may need to be inflated several times in order for the narrowed area to open up sufficiently to improve the blood flow. The area will be viewed with specialized x-ray or other imaging devices to see if the artery has opened enough.
  The UltraScore Focused Force PTA balloon through the blood vessel to the narrowed area to be treated.

SUMMARY:
The objective of this study is to assess the clinical use of the Bard® UltraScore™ Focused Force PTA balloon in a heterogeneous patient population in a real world, on-label clinical application.

DETAILED DESCRIPTION:
The registry is a prospective, multi-center, single-arm, real-world study to assess the clinical use of the Bard® UltraScore™ Focused Force PTA balloon for the treatment of stenotic lesions of the superficial femoral artery (SFA), popliteal artery, and infra-popliteal arteries (posterior tibial, anterior tibial and peroneal arteries). Follow-up for all treated subjects will be performed at hospital discharge, 30 days, and 6 and 12 months post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must voluntarily sign and date the Informed Consent Form (ICF) prior to collection of study data or performance of study procedures.
2. Subject must be either a male or non-pregnant female ≥ 21 years of age with an expected lifespan sufficient to allow for completion of all study procedures.
3. Subject must be willing to comply with the protocol requirements, including the follow-up procedures.
4. Subject must have a target lesion (de novo lesion or prior failed treatment) that can be treated with the UltraScore™ Focused Force PTA balloon according to the Instructions for Use (IFU). Only a target lesion in the SFA, popliteal, or infra-popliteal arteries (posterior tibial, anterior tibial, or peroneal arteries) may be treated for this study.
5. Subject must have an Above the Knee (ATK) or Below the Knee (BTK) target lesion with at least one vessel run-off.
6. The target lesion must be able to be crossed using a guidewire (use of chronic total occlusion (CTO) or atherectomy is allowed).

Exclusion Criteria:

1. Subjects that are to receive one or more stents as adjunctive therapy at the target lesion (bail out stenting is allowed).
2. The subject has a single target lesion that involves both ATK and BTK arteries.
3. The subject has a target lesion in a previously placed stent or stent graft (in-stent restenosis).
4. The subject has a lesion, which in the opinion of the Investigator, would preclude safe use of the UltraScore™ Focused Force PTA balloon.
5. The subject has a flow limiting dissection at the target lesion prior to use of the UltraScore™ Focused Force PTA balloon.
6. The subject has acute limb ischemia.
7. The subject has been assessed Rutherford category 6.
8. The subject has a known allergy or sensitivity to contrast media, which cannot be adequately pre-medicated.
9. The subject has another medical condition or is currently participating in an investigational drug or another device study that, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include a maximum of 350 subjects at up to 45 U.S. sites. All subjects will have peripheral arterial disease (PAD; a stenotic lesion of the SFA, popliteal, or infra-popliteal arteries).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Walker, MD, Principal Investigator — Cardiovascular Institute of the South (CIS) Clinical Research Corporation; Robert Beasley, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Miguel Montero, MD, Principal Investigator — Baylor St. Luke's College of Medicine
Locations (31):
- United States (31):
  - St. Luke's Hospital- Phoenix, Phoenix, Arizona
  - Health One Denver Heart, Denver, Colorado
  - Mount Sinai Medical Center, Miami Beach, Florida
  - St. Joseph Hospital, Fort Wayne, Indiana
  - Community Hospital Munster Research Foundation, Munster, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Willis Knighton Medical Center, Bossier City, Louisiana
  - CIS Clinical Research Corporation, Lafayette, Louisiana
  - MedStar Health Research Institute, Annapolis, Maryland
  - Beth Israel Deaconess Medical Center, Inc, Boston, Massachusetts
  - Providence-Providence Park Hospital, Southfield, Michigan
  - SSM DePaul Health Center, Bridgeton, Missouri
  - St. Louis Univeristy, St Louis, Missouri
  - Methodist Health System, Omaha, Nebraska
  - Mount Sinai School of Medicine, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Montefiore Medical Center, The Bronx, New York
  - East Carolina University, Greenville, North Carolina
  - Rex Hospital, Inc, Raleigh, North Carolina
  - Coastal Surgery Specialists, Wilmington, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - US Cardiovascular Jefferson Hills, Jefferson Hills, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Vascular Access Solutions, Orangeburg, South Carolina
  - Stern Cardiovascular Foundation, Inc, Germantown, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Baylor St. Luke's Health College of Medicine, Houston, Texas
  - The Methodist Hospital Research Institute dba Houston Methodist Research Institute, Houston, Texas
  - Texas Tech University Health Science Center/University Medical Center, Lubbock, Texas
  - HSHS St. Vincent Hospital, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PTA-UltraScore Focused Force PTA Balloon: Treatment with the UltraScore Focused Force PTA balloon will be per the investigational site's standard of care and adhering to the IFU.
  PTA (UltraScore Focused Force PTA Balloon): Percutaneous Transluminal Angioplasty (PTA) will involve the insertion of a catheter into one of the femoral arteries. Once the catheter is in place, a tiny balloon on the end of the catheter will be inflated to press against the narrowing (or blockage) in the artery to try to open the blockage, and allow more blood to flow through the artery. The balloon may need to be inflated several times in order for the narrowed area to open up sufficiently to improve the blood flow. The area will be viewed with specialized x-ray or other imaging devices to see if the artery has opened enough.
  The UltraScore Focused Force PTA balloon through the blood vessel to the narrowed area to be treated.
Period: Overall Study
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Started | 350
Completed | 349 (denominator for the primary endpoint analysis which was achieved at the point of index surgery)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 120
  >=65 years | 230
Age, Continuous [Mean (Full Range); unit: years] | 70.2 [45 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 238
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 80
  White | 239
  More than one race | 14
  Unknown or Not Reported | 16
Region of Enrollment [Number; unit: participants]
  United States | 350

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieve Optimal PTA Results
Description: Optimal result is defined as ≤30% residual stenosis without major flow-limiting dissection, as measured by angiographic imaging. Major flow limiting dissections are classified by the National Heart, Lung, and Blood Institute (NHLBI) as Grade D (Spiral luminal filling defects), Grade E (Appearance of new and persistent filling defects with reduced flow), and Grade F (Total occlusion without distal flow).
Time Frame: Index procedure (Day 0); approximate duration of procedure is 90 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 349
Participants | 254

2. Primary Outcome: Number of Participants With Technical Success of Use of UltraScore™ Focused Force PTA Balloon
Description: Technical success is determined subjectively by the investigator according to delivery location of the study device relative to the target lesion, as assessed by angiographic imaging, and inflation without movement.
Time Frame: Index procedure (Day 0); approximate duration of procedure is 90 minutes.
Population: Number of participants treated with Ultrascore.
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 350
Participants | 350

3. Secondary Outcome: Number of Participants With Bail-out Stenting Due to Dissection
Description: Number of participants who needed stent placement for abrupt or threatened artery closure caused by arterial dissection immediately following index procedure.
Time Frame: Index procedure (Day 0); approximate duration of procedure is 90 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 350
Participants | 14

4. Secondary Outcome: Number of Participants That Did Not Have a Target Lesion Revascularization (TLR).
Description: TLR is defined as a revascularization procedure (e.g. PTA, stenting, surgical bypass, etc.) in target vessel after the index procedure
Time Frame: 30 days post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 343
Participants | 343

5. Secondary Outcome: Number of Participants That Did Not Have a Target Lesion Revascularization (TLR).
Description: as for outcome 4
Time Frame: 6 months post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 307
Participants | 287

6. Secondary Outcome: Number of Participants That Did Not Have a Target Lesion Revascularization (TLR).
Description: as for outcome 4
Time Frame: 12 months post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 263
Participants | 232

7. Secondary Outcome: Number of Participants That Did Not Have a Major Amputation of the Target Limb
Description: Major amputation is defined as above the ankle amputation
Time Frame: 30 days post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 346
Participants | 337

8. Secondary Outcome: Number of Participants That Did Not Have a Major Amputation of the Target Limb
Description: Major amputation is defined as above the ankle amputation
Time Frame: 6 months post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 320
Participants | 303

9. Secondary Outcome: Number of Participants That Did Not Have a Major Amputation of the Target Limb
Description: Major amputation is defined as above the ankle amputation
Time Frame: 12 months post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 271
Participants | 253

10. Secondary Outcome: Number of Participants That Had Improved Clinical Measures From Baseline (ABI)
Description: Resting ankle brachial index (ABI) for chronic limb ischemia measurements will be assessed clinically at follow-up and compared with baseline. ABI measurements: Mild to moderate if the ABI is between 0.4 and 0.9, and an ABI less than 0.40 is suggestive of severe PAD [19]. An ABI value greater than 1.3 is also considered abnormal, suggestive of non-compressible vessels.
Time Frame: 30 days post-index procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 249
score on a scale | 0.988 (0.1875)

11. Secondary Outcome: Number of Participants That Had Improved Clinical Measures From Baseline (ABI)
Description: as for outcome 10
Time Frame: 6 months post-index procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 191
score on a scale | 0.927 (0.2188)

12. Secondary Outcome: Number of Participants That Had Improved Clinical Measures From Baseline (ABI)
Description: as for outcome 10
Time Frame: 12 months post-index procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 178
score on a scale | 0.952 (0.2450)

13. Secondary Outcome: Number of Participants That Had Improved Clinical Measures From Baseline (Rutherford Classification)
Description: Rutherford classification (RC):
  0 Asymptomatic: documented peripheral arterial disease, without symptoms of claudication or ischemic pain
  1. Mild claudication: ischemic limb muscle pain that does not limit walking, or limits walking only after >2 blocks (>600 feet, or 2 football fields)
  2. Moderate claudication: ischemic limb muscle pain that limits walking to 1-2 blocks (300-600 feet, or 1-2 football fields)
  3. Severe claudication: ischemic limb muscle pain that limits walking to <1 block (<300 feet, or 1 football field)
  4. Ischemic rest pain: pain in the distal foot at rest felt to be due to limited arterial perfusion
  5. Minor tissue loss: non-healing ischemic ulcer(s) on distal leg, or focal gangrene with diffuse pedal ischemia
  6. Major tissue loss: ischemic gangrene extending above TM level, functional foot no longer salvageable without extensive resvascularization efforts
Time Frame: 30 days post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 301
Participants
  RC 0 | 142
  RC 1 | 57
  RC 2 | 32
  RC 3 | 14
  RC 4 | 11
  RC 5 | 43
  RC 6 | 2

14. Secondary Outcome: Number of Participants That Had Improved Clinical Measures From Baseline (Rutherford Classification)
Description: as for outcome 13
Time Frame: 6 months post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 228
Participants
  RC 0 | 118
  RC 1 | 39
  RC 2 | 22
  RC 3 | 25
  RC 4 | 10
  RC 5 | 13
  RC 6 | 1

15. Secondary Outcome: Number of Participants That Had Improved Clinical Measures From Baseline (Rutherford Classification)
Description: as for outcome 13
Time Frame: 12 months post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 211
Participants
  RC 0 | 112
  RC 1 | 30
  RC 2 | 22
  RC 3 | 23
  RC 4 | 12
  RC 5 | 12
  RC 6 | 0

16. Secondary Outcome: Number of Participants That Had an Open (Patent) Target Vessel for Above the Knee (ATK) Subjects
Description: ATK subjects have a target lesion of the SFA or popliteal artery only. Primary patency (patent or open target vessel) is measured by duplex ultrasound (DUS) core lab; the core lab determines whether target vessel is patent/open.
Time Frame: 30 days post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 144
Participants | 137

17. Secondary Outcome: Number of Participants That Had an Open (Patent) Target Vessel for Above the Knee (ATK) Subjects
Description: as for outcome 16
Time Frame: 6 months post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 111
Participants | 89

18. Secondary Outcome: Number of Participants That Had an Open (Patent) Target Vessel for Above the Knee (ATK) Subjects
Description: as for outcome 16
Time Frame: 12 months post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
Number analyzed (Participants) | 104
Participants | 64

ADVERSE EVENTS:
Time Frame: 3 years and 7 months
Arm/Group | PTA-UltraScore Focused Force PTA Balloon
All-Cause Mortality (participants affected / at risk) | 32/350
Serious Adverse Events (participants affected / at risk) | 45/350
Other Adverse Events (participants affected / at risk) | 0/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTA-UltraScore Focused Force PTA Balloon (N=350)
Vascular disorders (Vascular disorders) | 44 (44) — Arteriovenous fistula Embolism arterial Femoral artery dissection Femoral artery perforation Peripheral artery dissection Vasospasm
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Peripheral arterial reocclusion (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT03193619/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03193619/SAP_001.pdf